CLINICAL TRIAL: NCT06302868
Title: Doxy.me VR vs. Telemental Health-Based Exposure Therapy
Brief Title: Telemedicine-Based Virtual Reality Clinic for the Treatment of Phobias
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 006215; R43MH129065 (NIH)
Record Dates: First submitted 2024-01-12; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Arachnophobia; Cynophobia; Ophidiophobia
Keywords: phobia; phobias; snakes; dogs; spiders
MeSH Terms: conditions — Arachnophobia; Zoophobia; Phobic Disorders | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine-based Virtual Reality Exposure Therapy (Active Comparator): This group will receive exposure therapy in a telemedicine-based Virtual Reality Clinic using virtual reality snakes, dogs, or spiders. The VR stimuli range from small to medium to large and have four activity levels: idle, calm, energetic, and aggressive.
  Interventions: Behavioral: Telemedicine-Based Virtual Reality Exposure Therapy
- Standard Telemedicine Exposure Therapy (Active Comparator): This group will receive exposure therapy via Doxy.me telemedicine platform using photos and videos of snakes, dogs, or spiders. The photo/video stimuli range from small to medium to large and have four activity levels: idle, calm, energetic, and aggressive.
  Interventions: Behavioral: Telemedicine Exposure Therapy Using Photos and Videos

INTERVENTIONS:
Behavioral: Telemedicine Exposure Therapy Using Photos and Videos — Participants will complete 12 60-minute exposure therapy sessions using photos/videos and progress to in vivo exposures.
  Arms: Standard Telemedicine Exposure Therapy
Behavioral: Telemedicine-Based Virtual Reality Exposure Therapy — Participants will complete 12 60-minute exposure therapy sessions in a Virtual Reality Clinic using Virtual Reality stimuli and progress to in vivo exposures.
  Arms: Telemedicine-based Virtual Reality Exposure Therapy

SUMMARY:
The purpose of this study is to assess the feasibility of conducting a randomized controlled efficacy trial comparing the delivery of exposure therapy via a telemedicine-based virtual reality clinic (Doxy.me VR) vs. standard telemental health (TMH) to adults with intense fear of dogs, snakes, and/or spiders. The secondary purpose is to preliminarily examine the efficacy of using Doxy.me VR vs. TMH in reducing phobia severity.

DETAILED DESCRIPTION:
This study aims to assess the feasibility of conducting a randomized controlled efficacy trial comparing the delivery of exposure therapy via a telemedicine-based virtual reality clinic (Doxy.me VR) vs. standard telemental health (TMH) to adults with intense fear of dogs, snakes, and/or spiders. This study will use feasibility randomized controlled efficacy trial design. This single-site trial will include up to 60 adults with self-reported fear of dogs, snakes, and/or spiders who will be randomly assigned via the REDCap Randomization Module using a 1:1 allocation ratio to receive 12 sessions of exposure therapy over the course of 3 months via standard telemental health (TMH; n=15) vs. Doxy.me VR (n=15), a telemedicine-based virtual reality clinic.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Is an adult ≥ 18 years old
2. Has a self-reported fear of dogs, snakes, and/or spiders
3. Indicates Subthreshold or Present Specific Phobia symptoms as determined by the study therapist via administration of the Diagnostic Assessment Research Tool (DART) Specific Phobia Module
4. Has access to the internet AND a computer OR smartphone with video conferencing capabilities
5. Will reside in the state of Florida for the duration of the study

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Is participating in ongoing mental health therapy from a non-study therapist
2. Has had changes to psychotropic medication use within six weeks preceding enrollment in the trial
3. Reports active suicidal and/or homicidal intent or plan as determined by the study therapist via administration of the Diagnostic Assessment Research Tool (DART) Risk Assessment Module
4. Reports active auditory, visual, and/or tactile hallucinations via the Diagnostic Assessment Research Tool (DART) Psychosis Module screening question
5. Reports a history of epilepsy or seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Phobia symptom severity | 3 Month Follow-Up
  The Severity Measure for Specific Phobia (SMSP) will be used to assess changes in phobia symptom severity at the 3 Month Follow-Up.
  Each item on the measure is rated on a 5-point scale (0=Never; 1=Occasionally; 2=Half of the time; 3=Most of the time, and 4=All of the time). The total score can range from 0 to 40 with higher scores indicating greater severity of specific phobia. The clinician will use an average total score, which reduces the overall score to a 5-point scale, which allows the clinician to think of the severity of the individual's specific phobia in terms of none (0), mild (1), moderate (2), severe (3), or extreme (4).

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Bunnell, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuler KR, Ong T, Welch BM, Craggs JG, Bunnell BE. Examining a Telemedicine-Based Virtual Reality Clinic in Treating Adults With Specific Phobia: Protocol for a Feasibility Randomized Controlled Efficacy Trial. JMIR Res Protoc. 2025 Apr 10;14:e65770. doi: 10.2196/65770. PMID 40209221

DOCUMENTS (2):
  • Study Protocol (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT06302868/Prot_000.pdf
  • Informed Consent Form (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT06302868/ICF_001.pdf